CLINICAL TRIAL: NCT01430403
Title: Preventative Omalizumab or Step-up Therapy for Severe Fall Exacerbations (ICAC-20)
Brief Title: Preventative Omalizumab or Step-up Therapy for Severe Fall Exacerbations
Acronym: PROSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ICAC-20
Record Dates: First submitted 2011-09-01; First posted 2011-09-08 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: persistent allergic asthma; asthma exacerbations reduction; Xolair® (omalizumab); Flovent® Diskus® (fluticasone); placebo; inhaled corticosteroid therapy; anti-immunoglobulin E therapy; anti-IgE therapy
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Omalizumab (Experimental): Participants receive active omalizumab (Xolair®) injections and a placebo Flovent® Diskus® (fluticasone) inhaler. Each participant will receive omalizumab (Xolair®) subcutaneous injections at minimum dose of 0.016 mg/kg/IgE (immunoglobulin E) [IU/mL] every 2 or 4 weeks during the 4-5 months treatment period. In addition, all participants receive standardized specialist asthma care.
  Interventions: Biological: Omalizumab; Biological: Placebo fluticasone
- Inhaled Corticosteroid Boost Therapy (ICS) (Experimental): Participants in this group, the Inhaled Corticosteroid (ICS) boost arm, receive active ICS and placebo omalizumab (Xolair®) injections. Self-administered fluticasone (Flovent ® Diskus®) inhalers sufficient to deliver the required 200 mcg or 500 mcg daily boost of fluticasone will be used. In addition, all participants receive standardized specialist asthma care.
  Interventions: Drug: Inhaled Corticosteroid Boost Therapy (ICS); Biological: Placebo omalizumab
- Placebo (Placebo Comparator): The placebo group receive placebo omalizumab (Xolair®) injections and placebo Flovent® Diskus® (fluticasone) inhaler. In addition, all participants receive standardized specialist asthma care.
  Interventions: Biological: Placebo omalizumab; Biological: Placebo fluticasone

INTERVENTIONS:
Biological: Omalizumab — Participants received active omalizumab (Xolair(R)) injections and a placebo inhaler. Each participant received omalizumab (Xolair(R)) subcutaneous injections at minimum dose of 0.016 mg/kg/IgE (immunoglobulin E) [IU/mL] every 2 or 4 weeks during the 4-5 months treatment period. All participants received standardized specialist asthma care.
  Other Names: Xolair®
  Arms: Omalizumab
Drug: Inhaled Corticosteroid Boost Therapy (ICS) — Self-administered fluticasone (Flovent ® Diskus®) inhalers sufficient to deliver the required 200 mcg or 500 mcg daily boost of fluticasone. All participants will receive standardized specialist asthma care.
  Other Names: Flovent® Diskus®
  Arms: Inhaled Corticosteroid Boost Therapy (ICS)
Biological: Placebo omalizumab — Placebo was administered subcutaneously every 2 or 4 weeks over a period of 4 to 5 months. Doses (mg) and dosing frequency were determined by serum total immunoglobulin E (IgE) level (IU/mL) and body weight (kg). Also, participants continued with their conventional asthma therapy according to the National Asthma Education and Prevention Program (NAEPP, 2007) guidelines, under the management of an asthma specialist health care provider.
  Other Names: Placebo Xolair®
  Arms: Inhaled Corticosteroid Boost Therapy (ICS); Placebo
Biological: Placebo fluticasone — Self-administered placebo fluticasone (placebo Flovent ® Diskus®) inhalers identical in dose and guidance as active fluticasone. All participants will receive standardized specialist asthma care.
  Other Names: Placebo Flovent® Diskus®
  Arms: Omalizumab; Placebo

SUMMARY:
The purpose of this trial is to compare the efficacy of 4 to 5 months of three treatments - omalizumab, corticosteroid therapy boost, and placebo - in reducing fall exacerbations in inner-city children and adolescents with allergic persistent asthma when initiated approximately 4 -6 weeks prior to the start of the first day of each participant's school year.

DETAILED DESCRIPTION:
While the increase in the prevalence of asthma has abated, levels of asthma morbidity and mortality remain near record highs. An asthma exacerbation is a major factor contributing to morbidity, and even mortality in patients with asthma. Although current approaches to treatment have reduced these risks, asthma exacerbations are major problems for inner-city patients and their families, and prevention of these events continues to be a significant challenge. In children with asthma, there are predictable seasonal epidemics of exacerbations, especially during the fall season, otherwise known as the "September epidemic."

ELIGIBILITY:
Inclusion Criteria :

* Combined body weight (as measured at the screening visit) and total serum IgE level (as measured within 3 months of the screening visit) suitable for omalizumab (Xolair®) dosing;
* A diagnosis of asthma by a clinician made more than 1 year prior to recruitment; participants who received an asthma diagnosis by a clinician less than 1 year prior to recruitment must report that their respiratory symptoms were present for more than 1 year prior to recruitment;
* Having a requirement for at least 100 mcg fluticasone 100 mcg twice a day or equivalent at the Assumption of Care Visit AND who meet at least one of the following criteria:

  i. ≥1 asthma-related exacerbations, separated by at least two weeks, requiring treatment with a systemic corticosteroid course in the previous 12 months ii. ≥1 asthma-related overnight hospitalizations in the past 12 months.
* A positive prick skin-test to at least one perennial allergen (i.e. dust mite, cockroach, mold, cat, dog, rat, mouse) documented at the screening visit or at a ICAC study visit within 12 months of the screening visit;
* Primary place of residence is in one of the pre-selected recruitment census tracts;
* Able to perform spirometry;
* Parent or legal guardian is willing to sign the written informed consent (age appropriate) prior to initiation of any study procedure;
* Willing to sign the assent form, if age appropriate;
* A history of chickenpox or receipt of the chickenpox vaccine;
* Insurance which covers costs of medications; and
* Have not used and do not plan to restart any of the following medications in the 7 days prior to the first visit: tricyclic antidepressants, ketaconazole, or beta adrenergic blocker drugs (oral and/or topical).

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for enrollment but may be reassessed:

* Assigned to a treatment of less than 100 mcg fluticasone twice a day or equivalent at the Assumption of Care Visit;
* Pregnant or lactating. Females of child-bearing potential (post-menarche) must be abstinent or use a medically acceptable birth control method throughout the study (e.g. oral, subcutaneous, mechanical, or surgical contraception);
* Clinically significant laboratory abnormalities (not associated with the study indication) at the screening visit;
* Platelet count less than 100 x 10^9/L at the screening visit;
* Currently participating in another asthma-related pharmaceutical study or intervention study or who have participated in another asthma-related pharmaceutical study or intervention study in the month prior to Recruitment;
* Living with a foster parent: exception -not applicable if participant is able to provide consent;
* Does not have access to a phone (needed for scheduling appointments);
* Plan(s) to move from the area during the study period;
* Has previously been treated with omalizumab (Xolair®) within 1 year of recruitment;
* Currently receiving or has received hyposensitization therapy to any allergen in the past year prior to recruitment;
* Has received hyposensitization therapy to dust mite, Alternaria or cockroach for ≥ 6 months in the past 3 years prior to Recruitment;
* Has experienced a life-threatening asthma exacerbation in the last 2 years requiring intubation, mechanical ventilation, or resulting in a hypoxic seizure;
* Home-schooled or in year round school;
* Are currently taking or who have taken any of the following medications within 4 weeks of the Screening Visit: monoamine oxidase inhibitors (phenelzine, tranylcypromine); tricyclic and tetracyclic antidepressants; beta adrenergic blocker drugs (both oral and topical); anticonvulsants(carbamazepine, phenobarbital, phenytoin, mephobarbital, primidone,ethosuximide, methsuximide, felbamate, gabapentin, lamotrigine, levetiracetam, oxcarbazepine, tiagabine, topiramate, valproic acid, divalproex sodium, zonisamide); protease inhibitors(ritonavir, indinavir, nelfinavir); calcium channel blockers (verapamil, diltiazem); modafinil; tamoxifen; non-nucleoside reverse transcriptase inhibitors; macrolide antibiotics*(erythromycin, clarithromycin, dirithromycin, troleandomycin); chloramphenicol; nefazodone; aprepitant; St. John's Wort (hypericum); Rifampin*; Azole antifungals* (ketoconazole, fluconazole,itraconazole); Sibutramine*; bergamottin* (constituent of grapefruit juice).*may be rescreened if this therapy is short-lived;
* Will not allow the study clinician, an asthma specialist, to manage their disease for the duration of the study or who are not willing to change their asthma medications to follow the protocol.

Participants who meet any of the following criteria are not eligible for assumption of care and may not be reassessed except where noted:

* A current severe hypersensitivity to milk;
* Individuals who were enrolled in the previous ICAC trial, Inner-City Anti-IgE Therapy for Asthma (ICATA,ICAC-NCT00377572);
* Individuals who have any medical illnesses that in the opinion of the investigators would a.) increase the risk the subject would incur by participating in the study; b.) interfere with the measured outcomes of the study; or c.) interfere with the performance of the study procedures. Examples of such diseases are: cystic fibrosis, bronchiectasis, type 1 diabetes, hemophilia, Von Willebrand disease, sickle cell disease, cerebral palsy, rheumatoid arthritis, lupus, psoriasis, hyperimmunoglobulin E syndrome, parasite infections, Wiskott-Aldrich Syndrome or allergic bronchopulmonary aspergillosis.
* Known hypersensitivity to any ingredients, including excipients (sucrose, histidine, polysorbate 20) of the study medication or drugs related to omalizumab (e.g. monoclonal antibodies, polyclonal gamma globulin) or fluticasone;
* Currently have diagnosed cancer, are currently being investigated for possible cancer, or who have a history of cancer;
* Do not primarily speak English (or Spanish at centers with Spanish speaking staff)
* The participant's caretaker does not primarily speak English (or Spanish at centers with Spanish speaking staff); not applicable if participant is able to provide consent.
* A history of severe(grade 3) anaphylactoid or anaphylactic reaction(s).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 478 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Szefler, MD, Study Chair — National Jewish Health; Stephen Teach, MD, MPH, Study Chair — Children's National Research Institute
Locations (8):
- United States (8):
  - National Jewish Health, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Department of Allergy, Chicago, Illinois
  - Boston University School of Medicine, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Result] Teach SJ, Gill MA, Togias A, Sorkness CA, Arbes SJ Jr, Calatroni A, Wildfire JJ, Gergen PJ, Cohen RT, Pongracic JA, Kercsmar CM, Khurana Hershey GK, Gruchalla RS, Liu AH, Zoratti EM, Kattan M, Grindle KA, Gern JE, Busse WW, Szefler SJ. Preseasonal treatment with either omalizumab or an inhaled corticosteroid boost to prevent fall asthma exacerbations. J Allergy Clin Immunol. 2015 Dec;136(6):1476-1485. doi: 10.1016/j.jaci.2015.09.008. Epub 2015 Oct 27. PMID 26518090
- [Derived] Szefler SJ, Casale TB, Haselkorn T, Yoo B, Ortiz B, Kattan M, Busse WW. Treatment Benefit with Omalizumab in Children by Indicators of Asthma Severity. J Allergy Clin Immunol Pract. 2020 Sep;8(8):2673-2680.e3. doi: 10.1016/j.jaip.2020.03.033. Epub 2020 Apr 13. PMID 32298853
- [Derived] Esquivel A, Busse WW, Calatroni A, Togias AG, Grindle KG, Bochkov YA, Gruchalla RS, Kattan M, Kercsmar CM, Khurana Hershey G, Kim H, Lebeau P, Liu AH, Szefler SJ, Teach SJ, West JB, Wildfire J, Pongracic JA, Gern JE. Effects of Omalizumab on Rhinovirus Infections, Illnesses, and Exacerbations of Asthma. Am J Respir Crit Care Med. 2017 Oct 15;196(8):985-992. doi: 10.1164/rccm.201701-0120OC. PMID 28608756
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/research/role
- See also: Inner City Asthma Consortium (ICAC) Description and Goals — http://www.niaid.nih.gov/topics/asthma/research/Pages/innerCity.aspx#icac

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight National Institute of Allergy and Infectious Diseases (NIAID) Inner-City Asthma Consortium (ICAC) sites in the United States recruited the targeted number of study participants who fulfilled entry criteria. Recruitment occurred September 2011 to March 2014.
Groups:
- Inhaled Corticosteroid Boost Therapy (ICS): Participants in the Inhaled Corticosteroid (ICS) boost arm received active ICS and placebo injections of omalizumab (Xolair(R)). Self-administered fluticasone (Flovent (R) Diskus) inhalers sufficient to deliver the required 200 mcg or 500 mcg daily boost of fluticasone were used. All participants received standardized specialist asthma care.
- Placebo: Participants in the placebo group received placebo injection and placebo inhaler. All participants received standardized specialist asthma care.
Period: Overall Study
Arm/Group | Omalizumab | Inhaled Corticosteroid Boost Therapy (ICS) | Placebo
Started | 259 (Intent-to-treat) | 130 (Intent-to-treat) | 89 (Intent-to-treat)
Completed | 242 | 121 | 81
Not Completed | 17 | 9 | 8
Not completed — Lost to Follow-up | 5 | 5 | 3
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 3 | 2
Not completed — Withdrawal by Subject | 9 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Inhaled Corticosteroid Boost Therapy (ICS) | Placebo | Total
Number analyzed (Participants) | 259 | 130 | 89 | 478
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 259 | 130 | 89 | 478
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Customized [Number; unit: participants]
  6-11 years | 190 | 102 | 67 | 359
  12-17 years | 69 | 28 | 22 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 60 | 30 | 175
  Male | 174 | 70 | 59 | 303
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 88 | 43 | 30 | 161
  Not Hispanic or Latino | 171 | 87 | 59 | 317
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 2 | 9
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 152 | 82 | 57 | 291
  White | 37 | 18 | 9 | 64
  More than one race | 27 | 12 | 9 | 48
  Unknown or Not Reported | 36 | 16 | 11 | 63
Region of Enrollment [Number; unit: participants]
  United States | 259 | 130 | 89 | 478

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of One or More Asthma Exacerbations (All Treatment Steps [Steps 2-5])
Description: Asthma exacerbation defined as a prescribed course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant or a hospitalization during the fall outcome period (90 day period beginning on the first day of the participant's school year) to prevent a serious asthma outcome. If a participant initiates and completes a course of systemic steroids without clinician involvement, this course will be counted only if it meets the following minimum dosage: prednisone, prednisolone, or methylprednisolone at ≥ 20mg per day for 3 of any 5 consecutive days; or dexamethasone at ≥10mg per day for ≥1 day. Odds ratio comparing Placebo and Omalizumab arms across all treatment steps (Steps 2-5).
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Number; unit: Percent of adjusted prevalence
Groups:
- Treatment Steps 2-5: Omalizumab: Participants on the omalizumab arm across all treatment steps (2-5) at randomization. Six treatment steps were established, consistent with report 3 of the National Asthma Education and Prevention Program guidelines to standardize prescribing patterns according to levels of asthma severity. Steps 1 and 2 apply to mild asthma, Step 3 to moderate asthma, and Steps 4 through 5 to severe asthma.
- Treatment Steps 2-5: Placebo: Participants on the placebo arm across all treatment steps (2-5) at randomization. Six treatment steps were established, consistent with report 3 of the National Asthma Education and Prevention Program guidelines to standardize prescribing patterns according to levels of asthma severity. Steps 1 and 2 apply to mild asthma, Step 3 to moderate asthma, and Steps 4 through 5 to severe asthma.
Arm/Group | Treatment Steps 2-5: Omalizumab | Treatment Steps 2-5: Placebo
Number analyzed (Participants) | 259 | 89
Percent of adjusted prevalence | 11.3 | 21.0
Statistical Analysis 1: Comparison: Treatment Steps 2-5: Omalizumab vs Treatment Steps 2-5: Placebo; Null hypothesis is that there is no difference between the arms. Power calculation is described in detail in the study protocol; Test type: Superiority or Other; p = 0.03, Odds Ratio; Adjusted for Site, dosing group and treatment step; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.25 to 0.92], Standard Error of Mean 0.331 — Placebo serves as the reference group. Values < 1 represent more exacerbations in the placebo arm

2. Primary Outcome: Occurrence of One or More Asthma Exacerbations (Treatment Steps 2-4)
Description: Asthma exacerbation defined as a prescription of a course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant or a hospitalization during the fall outcome period (90 day period beginning on the first day of the participant's school year) to prevent a serious asthma outcome. If a participant initiates and completes a course of systemic steroids without clinician involvement, this course will be counted only if it meets the following minimum dosage: prednisone, prednisolone, or methylprednisolone at ≥20mg per day for 3 of any 5 consecutive days; or dexamethasone at ≥10mg per day for ≥1 day. Odds ratio comparing Inhaled corticosteroid boost therapy (ICS) and Omalizumab arms at Treatment Steps 2-4.
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Number; unit: Percent of adjusted prevalence
Groups:
- Treatment Steps 2-4: Omalizumab: Participants on the omalizumab arm at Treatment Steps 2-4 at randomization. Six treatment steps were established, consistent with report 3 of the National Asthma Education and Prevention Program guidelines to standardize prescribing patterns according to levels of asthma severity. Steps 1 and 2 apply to mild asthma, Step 3 to moderate asthma, and Steps 4 through 5 to severe asthma.
- Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS): Participants on the ICS arm at Treatment Steps 2-4 at randomization. Six treatment steps were established, consistent with report 3 of the National Asthma Education and Prevention Program guidelines to standardize prescribing patterns according to levels of asthma severity. Steps 1 and 2 apply to mild asthma, Step 3 to moderate asthma, and Steps 4 through 5 to severe asthma.
Arm/Group | Treatment Steps 2-4: Omalizumab | Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS)
Number analyzed (Participants) | 121 | 130
Percent of adjusted prevalence | 8.4 | 11.1
Statistical Analysis 1: Comparison: Treatment Steps 2-4: Omalizumab vs Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.45, Odds Ratio; Adjusted for Site, dosing group and treatment step; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.33 to 1.64], Standard Error of Mean 0.41 — ICS Boost serves as the reference group. Values < 1 represent more exacerbations in the ICS arm

3. Secondary Outcome: Virus-induced Exacerbations as Measured by an Exacerbation That is Associated With a Virus Detected Using the Nasal Mucus Samples
Description: Asthma exacerbation:defined by a prescribed course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant or a hospitalization during the fall outcome period (90 day period beginning on the 1st day of the participant's school year) to prevent a serious asthma outcome. If a participant initiates and completes a course of systemic steroids without clinician involvement, this course will be counted only if it meets the following minimum dosage: prednisone, prednisolone, or methylprednisolone at ≥ 20mg per day for 3 of any 5 consecutive days; or dexamethasone at ≥ 10mg per day for ≥1 day. Exacerbations were then associated with viral respiratory infections based on nasal mucus samples collected monthly. Nasal mucus samples were categorized as having exacerbations or not having exacerbations. Participants could potentially be counted in each group, as participants could have samples with exacerbations and samples without exacerbations.
Time Frame: 90 Day outcome period
Population: Nasal mucus samples
Measure: Number; unit: Percent Samples with virus
Units Other Than Participants: Number of Samples Analyzed
Groups:
- Samples With Exacerbations: These nasal mucus samples were associated with an exacerbation (defined as a prescribed course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant or a hospitalization during the fall outcome period (90 day period beginning on the first day of the participant's school year) to prevent a serious asthma outcome. If a participant initiates and completes a course of systemic steroids without clinician involvement, this course will be counted only if it meets the following minimum dosage: prednisone, prednisolone, or methylprednisolone at >/= 20mg per day for 3 of any 5 consecutive days; or dexamethasone at >/= 10mg per day for >/= 1 day)
- Samples Without Exacerbations: These nasal mucus samples were not associated with an exacerbation (defined as a prescribed course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant or a hospitalization during the fall outcome period (90 day period beginning on the first day of the participant's school year) to prevent a serious asthma outcome. If a participant initiates and completes a course of systemic steroids without clinician involvement, this course will be counted only if it meets the following minimum dosage: prednisone, prednisolone, or methylprednisolone at >/= 20mg per day for 3 of any 5 consecutive days; or dexamethasone at >/= 10mg per day for >/= 1 day)
Arm/Group | Samples With Exacerbations | Samples Without Exacerbations
Number analyzed (Participants) | 67 | 462
Number analyzed (Number of Samples Analyzed) | 149 | 5061
Percent Samples with virus | 71.8 | 40.4
Statistical Analysis 1: Comparison: Samples With Exacerbations vs Samples Without Exacerbations; Test type: Superiority or Other; p < 0.01, Chi-squared; Odds Ratio (OR) = 3.53, 95% CI 2-sided [2.38 to 5.22] — Adjusted for site

4. Secondary Outcome: Severity of Asthma Symptoms Associated With a Viral Infection:Omalizumab vs. Placebo
Description: Severity asthma symptoms is defined as the highest value among the following 3 variables: number of days with wheezing, tightness in the chest, or cough; number of nights with disturbed sleep as a result of asthma; and number of days on which a participant had to slow down or discontinue play/physical activities over a two week period associated with a viral infection. This outcome looks at the effect by group on number of days with asthma symptoms and infections. The hypothesis behind this outcome measure is that omalizumab will change virology; thus, the the intent of this measure was to assess the comparator group of placebo against omalizumab
Time Frame: 90 Day outcome period
Population: The pre-specified intent for Outcome Measure: analysis inclusion limited to the Omalizumab and Placebo Groups.
  Analysis: intent-to-treat (with available data).
Measure: Mean (Standard Error); unit: Maximum Symptoms Days
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 259 | 89
Maximum Symptoms Days | 1.2 (0.09) | 1.8 (0.23)
Statistical Analysis 1: Comparison: Omalizumab; Test type: Superiority or Other; p = 0.94, F-Test; Linear Regression = 0.004, 95% CI 2-sided [-0.10 to 0.11]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = 0.33, F-Test; Linear Regression = -0.13, 95% CI 2-sided [-0.40 to 0.13]

5. Secondary Outcome: Number of Exacerbations Evaluated Monthly With Viral Respiratory Infections: Omalizumab vs. Placebo
Description: Asthma exacerbation is defined as a prescribed course of systemic steroids by a clinician or initiation of a course of systemic steroids by a participant or a hospitalization during the fall outcome period (90 day period beginning on the first day of the participant's school year) to prevent a serious asthma outcome. If a participant initiates and completes a course of systemic steroids without clinician involvement, this course will be counted only if it meets the following minimum dosage: prednisone, prednisolone, or methylprednisolone at ≥20mg per day for 3 of any 5 consecutive days; or dexamethasone at ≥10mg per day for ≥1 day. The hypothesis behind this outcome measure is that omalizumab will change virology; thus, the intent of this measure was to assess the comparator group of placebo against omalizumab.
Time Frame: 90 Day outcome period
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Total Number of Viral Infections
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 163 | 65
Total Number of Viral Infections | 5.6 (0.19) | 5.8 (0.13)
Statistical Analysis 1: Comparison: Omalizumab; Test type: Superiority or Other; p = 0.552, Chi-squared; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.87 to 1.31]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = 0.37, Chi-squared; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.87 to 1.44]

6. Secondary Outcome: Composite Asthma Severity Index (CASI), Treatment Steps 2-5: Omalizumab vs. Placebo
Description: CASI scores include 5 domains: day symptoms and albuterol use, night symptoms and albuterol use, controller treatment, lung function measures, and exacerbations. To calculate CASI, the 5 domain scores are summed to determine a final score, which can range from 0 to 20, with 0 being no severity of asthma and 20 being extremely severe asthma.
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: CASI Score
Arm/Group | Treatment Steps 2-5: Omalizumab | Treatment Steps 2-5: Placebo
Number analyzed (Participants) | 259 | 89
CASI Score | 4.9 (0.15) | 5.5 (0.27)
Statistical Analysis 1: Comparison: Treatment Steps 2-5: Omalizumab vs Treatment Steps 2-5: Placebo; Test type: Superiority or Other; p = 0.09, Regression, Linear; Adjustments for randomization CASI, site, dosing group and treatment group step (2-4 as one step and 5 separately); Mean Difference (Net) = -0.52, 95% CI 2-sided [-1.11 to 0.07], Standard Error of Mean 0.30

7. Secondary Outcome: Composite Asthma Severity Index (CASI), Treatment Steps 2-4: Omalizumab vs. ICS
Description: as for outcome 6
Time Frame: 90 Day outcome period
Population: Intent-to-treat with available CASI scores
Measure: Mean (Standard Error); unit: CASI Score
Arm/Group | Treatment Steps 2-4: Omalizumab | Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS)
Number analyzed (Participants) | 82 | 101
CASI Score | 4.6 (0.23) | 4.8 (0.24)
Statistical Analysis 1: Comparison: Treatment Steps 2-4: Omalizumab vs Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS); Test type: Superiority or Other; p = 0.39, Regression, Linear; Adjustments for randomization CASI, site and dosing group; Mean Difference (Net) = -0.26, 95% CI 2-sided [-0.86 to 0.34], Standard Error of Mean 0.30

8. Secondary Outcome: Spirometry Measurements: Forced Expiratory Volume in 1 Second (FEV1) % Predicted, Treatment Steps 2-5:Omalizumab vs. Placebo
Description: FEV1 is air volume exhaled in 1 second during spirometry. Asthma severity classification for trial: mild--pre-bronchodilator FEV1 ≥ 80% predicted requiring no/ low-moderate dose of inhaled glucocorticoids; moderate--pre-bronchodilator FEV1 <80% predicted requiring no/ low-moderate dose of inhaled glucocorticoids; severe--requiring high-dose inhaled glucocorticoids with/without continuous/near continuous oral glucocorticoids, or uncontrolled despite treatment. FEV1 percent of predicted value is FEV1 converted to a percentage of normal, based on height, weight, and race.
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: percent predicted FEV1
Arm/Group | Treatment Steps 2-5: Omalizumab | Treatment Steps 2-5: Placebo
Number analyzed (Participants) | 259 | 89
percent predicted FEV1 | 92.2 (0.79) | 92.5 (1.38)
Statistical Analysis 1: Comparison: Treatment Steps 2-5: Omalizumab vs Treatment Steps 2-5: Placebo; Test type: Superiority or Other; p = 0.84, Regression, Linear; Adjustments for randomization FEV1 % predicted, site, dosing group and treatment group step (2-4 as one step and 5 separately); Mean Difference (Net) = -0.32, 95% CI 2-sided [-3.42 to 2.78], Standard Error of Mean 1.58

9. Secondary Outcome: Spirometry Measurements: Forced Expiratory Volume in 1 Second (FEV1) % Predicted , Treatment Steps 2-4: Omalizumab vs. ICS
Description: as for outcome 8
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: percent predicted FEV1
Arm/Group | Treatment Steps 2-4: Omalizumab | Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS)
Number analyzed (Participants) | 121 | 130
percent predicted FEV1 | 93.2 (1.15) | 90.8 (1.16)
Statistical Analysis 1: Comparison: Treatment Steps 2-4: Omalizumab vs Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS); Test type: Superiority or Other; p = 0.14, Regression, Linear; Adjustments for randomization FEV1 % predicted, site and dosing group; Median Difference (Net) = 2.37, 95% CI 2-sided [-0.76 to 5.51], Standard Error of Mean 1.59

10. Secondary Outcome: Spirometry Measurements: FEV1:FVCx100, Treatment Steps 2-5: Omalizumab vs. Placebo
Description: The FEV1 (forced expiratory volume 1))/ FVC (forced vital capacity) ratio is used to evaluate airways obstructions since pure restrictive ventilatory defects cause an equal reduction in the FEV1 and the FVC. An FEV1/FVC ratio below 80% indicates airflow obstruction. Normal FEV1/FVC: 8 - 19 years of age=85%.
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: percent FEV1/FVC ratio
Arm/Group | Treatment Steps 2-5: Omalizumab | Treatment Steps 2-5: Placebo
Number analyzed (Participants) | 259 | 89
percent FEV1/FVC ratio | 78.6 (0.44) | 78.4 (0.78)
Statistical Analysis 1: Comparison: Treatment Steps 2-5: Omalizumab vs Treatment Steps 2-5: Placebo; Test type: Superiority or Other; p = 0.78, Regression, Linear; Adjustments for randomization FEV1:FVCx100, site, dosing group and treatment group step (2-4 as one step and 5 separately); Mean Difference (Net) = 0.25, 95% CI 2-sided [-1.49 to 1.99], Standard Error of Mean 0.89

11. Secondary Outcome: Spirometry Measurements: FEV1:FVCx100, Treatment Steps 2-4: Omalizumab vs. ICS
Description: as for outcome 10
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: percent FEV1/FVC ratio
Arm/Group | Treatment Steps 2-4: Omalizumab | Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS)
Number analyzed (Participants) | 121 | 130
percent FEV1/FVC ratio | 79.1 (0.64) | 77.9 (0.65)
Statistical Analysis 1: Comparison: Treatment Steps 2-4: Omalizumab vs Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS); Test type: Superiority or Other; p = 0.20, Regression, Linear; Adjustments for randomization FEV1:FVCx100, site and dosing group; Mean Difference (Net) = 1.15, 95% CI 2-sided [-0.61 to 2.91], Standard Error of Mean 0.89

12. Secondary Outcome: Asthma Control Test Scores: Asthma Control Test (ACT), Treatment Steps 2-5: Omalizumab vs. Placebo
Description: Outcome measure description: The Asthma Control Test (ACT) is a validated tool to assess asthma control (over the last 4 weeks) in patients ≥12 yrs old. It is comprised of 5 questions assessing symptoms, use of rescue medications, and the impact of asthma on everyday functioning. All questions are scored on a 5-point Likert scale (higher score indicating better control). Total scores can range from 5-25. A score of ≤19 is indicative of not well-controlled asthma. The minimally important difference is 3 points.
Time Frame: 90 Day outcome period
Population: Intent-to-treat with available ACT scores
Measure: Mean (Standard Error); unit: ACT Score
Arm/Group | Treatment Steps 2-5: Omalizumab | Treatment Steps 2-5: Placebo
Number analyzed (Participants) | 95 | 22
ACT Score | 22.9 (0.19) | 21.8 (0.35)
Statistical Analysis 1: Comparison: Treatment Steps 2-5: Omalizumab vs Treatment Steps 2-5: Placebo; Test type: Superiority or Other; p = 0.006, Regression, Linear; Adjustments for randomization ACT, site, dosing group and treatment group step (2-4 as one step and 5 separately); Mean Difference (Net) = 1.11, 95% CI 2-sided [0.32 to 1.90], Standard Error of Mean 0.40

13. Secondary Outcome: Asthma Control Test Scores: Asthma Control Test (ACT), Treatment Steps 2-4: Omalizumab vs. ICS
Description: The Asthma Control Test (ACT) is a validated tool to assess asthma control (over the last 4 weeks) in patients ≥12 yrs old. It is comprised of 5 questions assessing symptoms, use of rescue medications, and the impact of asthma on everyday functioning. All questions are scored on a 5-point Likert scale (higher score indicating better control). Total scores can range from 5-25. A score of ≤19 is indicative of not well-controlled asthma. The minimally important difference is 3 points.
Time Frame: 90 Day outcome period
Population: Intent-to-treat with available ACT Scores
Measure: Mean (Standard Error); unit: ACT Score
Arm/Group | Treatment Steps 2-4: Omalizumab | Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS)
Number analyzed (Participants) | 39 | 29
ACT Score | 23.0 (0.26) | 22.9 (0.32)
Statistical Analysis 1: Comparison: Treatment Steps 2-4: Omalizumab vs Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS); Test type: Superiority or Other; p = 0.89, Regression, Linear; Adjustments for randomization ACT, site and dosing group; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.76 to 0.86], Standard Error of Mean 0.41

14. Secondary Outcome: Asthma Control Test Score: Child Asthma Control Test (C-ACT), Treatment Steps 2-5: Omalizumab vs. Placebo
Description: The Childhood Asthma Control Test (C-ACT) is a validated tool to assess overall asthma control (over the last 4 weeks) in patients ages 4 to 11 years. Scores can range from 0 to 27. A score of 19 or less is indicative of asthma that is not well controlled. The minimally important difference in C-ACT scores is not defined
Time Frame: 90 Day outcome period
Population: Intent-to-treat with available C-ACT Scores
Measure: Mean (Standard Error); unit: C-ACT Score
Arm/Group | Treatment Steps 2-5: Omalizumab | Treatment Steps 2-5: Placebo
Number analyzed (Participants) | 190 | 67
C-ACT Score | 23.2 (0.19) | 22.5 (0.31)
Statistical Analysis 1: Comparison: Treatment Steps 2-5: Omalizumab vs Treatment Steps 2-5: Placebo; Test type: Superiority or Other; p = 0.05, Regression, Linear; Adjustments for randomization C-ACT, site, dosing group and treatment group step (2-4 as one step and 5 separately); Mean Difference (Net) = 0.71, 95% CI 2-sided [0.00 to 1.41], Standard Error of Mean 0.36

15. Secondary Outcome: Asthma Control Test Score: Child Asthma Control Test (C-ACT), Treatment Steps 2-4: Omalizumab vs. ICS
Description: as for outcome 14
Time Frame: 90 Day outcome period
Population: Intent-to-treat with available C-ACT Scores
Measure: Mean (Standard Error); unit: C-ACT Score
Arm/Group | Treatment Steps 2-4: Omalizumab | Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS)
Number analyzed (Participants) | 82 | 101
C-ACT Score | 23.7 (0.29) | 23.1 (0.26)
Statistical Analysis 1: Comparison: Treatment Steps 2-4: Omalizumab vs Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS); Test type: Superiority or Other; p = 0.12, Regression, Linear; Adjustments for randomization C-ACT, site and dosing group; Mean Difference (Net) = 0.58, 95% CI 2-sided [-0.15 to 1.30], Standard Error of Mean 0.37

16. Secondary Outcome: Work Disruptions Due to Child's Asthma, Treatment Steps 2-5: Omalizumab vs. Placebo
Description: The ratio of the work hours missed due to child's asthma over the numbers of work hours in the past 14 days among caretakers working.
Time Frame: 90 Day outcome period
Population: Intent-to-treat with available data
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Treatment Steps 2-5: Omalizumab | Treatment Steps 2-5: Placebo
Number analyzed (Participants) | 136 | 41
Ratio | 0.003 (0.001) | 0.004 (0.003)
Statistical Analysis 1: Comparison: Treatment Steps 2-5: Omalizumab vs Treatment Steps 2-5: Placebo; Test type: Superiority or Other; p = 0.63, Negative Binomial Generalized Estimating; Adjustments for site, dosing group and treatment group step (2-4 as one step and 5 separately); Rate Ratio = 0.72, 95% CI 2-sided [0.19 to 0.72], Standard Error of Mean 0.68

17. Secondary Outcome: Work Disruptions Due to Child's Asthma, Treatment Steps 2-4: Omalizumab vs. ICS
Description: as for outcome 16
Time Frame: 90 Day outcome period
Population: Intent-to-treat with available data
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Treatment Steps 2-4: Omalizumab | Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS)
Number analyzed (Participants) | 59 | 75
Ratio | 0.003 (0.001) | 0.003 (0.001)
Statistical Analysis 1: Comparison: Treatment Steps 2-4: Omalizumab vs Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS); Test type: Superiority or Other; p = 0.99, Negative Binomial Generalized Estimating; Adjustments for site and dosing group; Ratio = 1.00, 95% CI 2-sided [0.29 to 3.46], Standard Error of Mean 0.63

18. Secondary Outcome: School Absences (Percent), Treatment Steps 2-5:Omalizumab vs. Placebo
Description: The ratio of the number of school days missed over the numbers of school days in session
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Treatment Steps 2-5: Omalizumab | Treatment Steps 2-5: Placebo
Number analyzed (Participants) | 259 | 89
Ratio | 1.2 (0.20) | 1.6 (0.47)
Statistical Analysis 1: Comparison: Treatment Steps 2-5: Omalizumab vs Treatment Steps 2-5: Placebo; Test type: Superiority or Other; p = 0.31, Negative Binomial Generalized Estimating; Adjustments for site, dosing group and treatment group step (2-4 as one step and 5 separately); Ratio = 0.72, 95% CI 2-sided [0.39 to 1.35], Standard Error of Mean 0.32

19. Secondary Outcome: School Absences (Percent), Treatment Steps 2-4: Omalizumab vs. ICS
Description: The ratio of the number of school days missed over the numbers of school days in session
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Treatment Steps 2-4: Omalizumab | Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS)
Number analyzed (Participants) | 121 | 130
Ratio | 0.9 (0.25) | 2.0 (0.63)
Statistical Analysis 1: Comparison: Treatment Steps 2-4: Omalizumab vs Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS); Test type: Superiority or Other; p = 0.06, Negative Binomial Generalized Estimating; Adjustments for site and dosing group; Ratio = 0.48, 95% CI 2-sided [0.23 to 1.02], Standard Error of Mean 0.39

20. Secondary Outcome: Percent Adherence to Asthma Medication, Treatment Steps 2-5: Omalizumab vs. Placebo
Description: Adherence to the study regimen and other asthma treatments, assessed as percent of expected dose taken, by means of study interviews and study physician corroboration.
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: percent adherence
Arm/Group | Treatment Steps 2-5: Omalizumab | Treatment Steps 2-5: Placebo
Number analyzed (Participants) | 259 | 89
percent adherence | 88.6 (0.77) | 88.8 (1.28)
Statistical Analysis 1: Comparison: Treatment Steps 2-5: Omalizumab vs Treatment Steps 2-5: Placebo; Test type: Superiority or Other; p = 0.90, Regression, Linear; Adjustments for site, dosing group and treatment group step (2-4 as one step and 5 separately); Mean Difference (Net) = -0.18, 95% CI 2-sided [-3.08 to 2.72], Standard Error of Mean 1.48

21. Secondary Outcome: Percent Adherence to Asthma Medication, Treatment Steps 2-4: Omalizumab vs. ICS
Description: as for outcome 20
Time Frame: 90 Day outcome period
Population: Intent-to-treat
Measure: Mean (Standard Error); unit: percent adherence
Arm/Group | Treatment Steps 2-4: Omalizumab | Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS)
Number analyzed (Participants) | 82 | 101
percent adherence | 88.4 (1.12) | 88.6 (1.08)
Statistical Analysis 1: Comparison: Treatment Steps 2-4: Omalizumab vs Treatment Steps 2-4:Inhaled Corticosteroid Boost Therapy (ICS); Test type: Superiority or Other; p = 0.86, Regression, Linear; Adjustments for site and dosing group; Mean Difference (Net) = -0.28, 95% CI 2-sided [-3.26 to 2.71], Standard Error of Mean 1.52

22. Secondary Outcome: Comparison of Home Allergen (Cockroach) Exposure and Asthma Exacerbations: Omalizumab Versus Placebo
Description: Residential environmental exposure to cockroach allergen of participants in the context of the risk of asthma exacerbations and effect of omalizumab versus placebo (control) on asthma exacerbations was explored. Presence of cockroach allergen in household dust samples was assessed. Exacerbation defined as: participant required either 1.)a prescribed course of systemic steroids by a clinician2.)initiation of a course of systemic steroids or 3.)a hospitalization during the fall outcome period (90 day period beginning on the first day of the participant's school year) to prevent a serious asthma outcome. In cases that a participant initiated and completed a course of systemic steroids without clinician involvement, the course was counted as an exacerbation only with fulfillment of the following minimum dosage: prednisone, prednisolone, or methylprednisolone at ≥20mg per day for 3 of any 5 consecutive days; or dexamethasone at ≥10mg per day for ≥1 day).
Time Frame: 90 Day outcome period
Population: Prespecified Outcome Measure: analysis limited to the Omalizumab and Placebo Groups.
  Analysis: intent-to-treat (with available data).
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 179 | 61
Participants
  Exposure to cockroach. No exacerbations.: number analyzed (Participants) | 156 | 46
  Exposure to cockroach. No exacerbations. | 37 | 18
  Exposure to cockroach. Exacerbations: number analyzed (Participants) | 23 | 15
  Exposure to cockroach. Exacerbations | 7 | 2
  No exposure to cockroach. No exacerbations.: number analyzed (Participants) | 156 | 46
  No exposure to cockroach. No exacerbations. | 119 | 28
  No exposure to cockroach. Exacerbations: number analyzed (Participants) | 23 | 15
  No exposure to cockroach. Exacerbations | 16 | 13

ADVERSE EVENTS:
Time Frame: Treatment initiation visit to end of study.
Description: Adverse events reported for intent-to-treat population from the period spanning the initial treatment visit to end of study (up to 90 days).
Arm/Group | Omalizumab | Inhaled Corticosteroid Boost Therapy (ICS) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/259 | 0/130 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/259 | 1/130 | 1/89
Other Adverse Events (participants affected / at risk) | 41/259 | 16/130 | 12/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (N=259) | Inhaled Corticosteroid Boost Therapy (ICS) (N=130) | Placebo (N=89)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (N=259) | Inhaled Corticosteroid Boost Therapy (ICS) (N=130) | Placebo (N=89)
Nasopharyngitis (Infections and infestations) | 10 (13) | 8 (9) | 3 (3)
Headache (Nervous system disorders) | 17 (18) | 4 (5) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 16 (16) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No